CLINICAL TRIAL: NCT01134809
Title: Does Surgical Stress Impair Skeletal Muscle Protein and Carbohydrate Metabolism?
Brief Title: Skeletal Muscle Wasting and Insulin Resistance Following Surgical Stress
Acronym: SIRSS
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 09106
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Insulin Resistance
Keywords: Major abdominal surgery
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Major abdominal surgery: Patients having major abdominal surgery
  Interventions: Procedure: Major abdominal surgery

INTERVENTIONS:
Procedure: Major abdominal surgery — All adult patients having major abdominal surgery

SUMMARY:
Background: Skeletal muscle wasting or decrease in muscle mass occurs as a result of alteration in the body's mechanisms to make or break muscle protein. In animal models, the pathway termed as 'ubiquitin-proteasome pathway' (UPP) is primarily responsible for the regulation of skeletal muscle protein loss in wasting conditions and during infection(sepsis). Skeletal muscle wasting is noticed in patients having major surgery due to the inflammatory reaction triggered by special group of proteins called cytokines (inflammatory proteins), resulting in reduced muscle strength, impaired capacity to fight infections, change in bowel function, increased clinical complications and prolonged recovery. Major surgery also leads to decreased sensitivity to hormone known as insulin, resulting in 'diabeteslike'state.

We hypothesize that susceptibility of patients undergoing major abdominal surgery, to skeletal muscle wasting and insulin resistance, is determined by stress response to surgery over time, leading to changes in the pathways that make or break muscle protein, namely the Akt/Foxo signalling and UPP. Therefore, the aim of this study is to establish the underlying mechanisms of skeletal muscle wasting and insulin resistance in patients undergoing major abdominal surgery.

DETAILED DESCRIPTION:
Experimental plan Fifteen adult patients undergoing major open elective abdominal surgery will be included in this nonrandomized study.

Objectives:

1. To study the expression proteins and metabolites involved in UPP mediated protein degradation, in blood and muscle biopsy samples.
2. To correlate the effects of surgery on the release of bacteria in blood from the bowel.

The analysis of the samples will include the following techniques, namely, RTPCR, ELISA, western blotting and metabolomics.

Establishing the association between these signaling mechanisms and expression of the individual proteins secondary to inflammation following surgery and infection would enable application of suitable therapeutic strategies that could reduce the inflammatory response to benefit all patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing major open elective gastrointestinal surgery lasting 3 hours or more will be eligible for the study.

Exclusion Criteria:

* Patients who are:

  1. undergoing emergency surgery
  2. suffering from chronic illness, (e.g. diabetes) or other debilitating diseases
  3. on long term anti-inflammatory drugs, (e.g. NSAIDS, Steroids, immunosuppressant)
  4. on long term antibiotics
  5. on statins
  6. on full therapeutic dose of anticoagulants, or aspirin > 325 mg/day, clopidogrel > 75 mg/day
  7. suffering from bleeding diathesis
  8. unable to give consent
  9. pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients having major abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
postoperative insulin resistance | First week following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dileep N Lobo, Professor, Study Chair — University of Notitngham
Locations (1):
- University Hospitals Nottingham Queen's Medical Centre, Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Derived] Atkins R, Constantin-Teodosiu D, Varadhan KK, Constantin D, Lobo DN, Greenhaff PL. Major elective abdominal surgery acutely impairs lower limb muscle pyruvate dehydrogenase complex activity and mitochondrial function. Clin Nutr. 2021 Mar;40(3):1046-1051. doi: 10.1016/j.clnu.2020.07.006. Epub 2020 Jul 14. PMID 32711950
- [Derived] Varadhan KK, Constantin-Teodosiu D, Constantin D, Greenhaff PL, Lobo DN. Inflammation-mediated muscle metabolic dysregulation local and remote to the site of major abdominal surgery. Clin Nutr. 2018 Dec;37(6 Pt A):2178-2185. doi: 10.1016/j.clnu.2017.10.020. Epub 2017 Nov 2. PMID 29129636